CLINICAL TRIAL: NCT02985775
Title: Evaluate the Safety and Efficacy of Preemptive Adoptive CMV-specific T Cells Infusion for Prevention of Refractory CMV Infection in Patients After Haploidentical Stem Cell Transplantation
Brief Title: Preemptive Therapy With CMV-specific T Cells Infusion to Prevent Refractory CMV Infection Post Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, MD,PHD, Study Principal Investigator, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016PHB153
Record Dates: First submitted 2016-11-28; First posted 2016-12-07 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: CMV Infection
Keywords: CMV-specific T cell; haploidentical stem cell transplantation; immunologic response; acute GVHD
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Donor-derived CMVpp65-specific T cells (Experimental): Intervention to be adminstered is about 1 million per kg CMVpp65-specific T cells infusion once acute GVHD ocurred post haploidentical transplantation.
  Interventions: Biological: Donor-derived CMVpp65-specific T cells

INTERVENTIONS:
Biological: Donor-derived CMVpp65-specific T cells — About 1 million per kg CMVpp65-specific T cells will be infused once acute GVHD ocurred post haploidentical transplantation.

SUMMARY:
Cytomegalovirus (CMV) infections remain an important cause of morbidity and mortality in allogeneic hematopoietic cell transplant (HSCT) recipients, especially in patients received haploidentical transplantation. During the past decades, prophylactic or preemptive treatment with antiviral drugs has significantly reduce the incidence of early-onset CMV infection. Unfortunately, prolonged antiviral treatment is associated with substantial toxicity and may delay recovery of virus specific immune responses, resulting in an increasing of late-onset CMV disease.

To date, adoptive immunotherapies have been developed as treatment alternatives to antiviral agents for CMV infection after HSCT. Studies have demonstrated that prophylactic or preemptive therapy with donor CMV-specific T cells can restore antiviral immunity and clear CMV viremia after transplantation. In this prospective clinical phase I/II trial, we propose to reconstitute antiviral immunity against CMV by preemptive transfer of CMV-specific T cells at an early time point after allogeneic stem cell transplantation. We also propose to demonstrate whether protect against CMV is associated with recovery of CMV-specific T cells.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) patients enrolled into this clinical trial are standard risk patients diagnosed with acute leukemia or myelodysplastic syndrome (MDS) and received haploidentical blood and marrow transplantation. When patients develop acute graft versus host disease (aGVHD), CMVpp65-specific T cells will be generated and transferred to the aGVHD controlled patients(patients who do not develop aGVHD are at low risk of refractory CMV infection, and are not include in treated group). Physical exams and blood tests will be performed -2w, -0d before and +1d, +2w, +4w, +8w, +12w, +24w after adoptive CMV-CTL transfusion. The end points were safety and clinical and immunologic response. Following time is 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Primary disease is leukemia or MDS.
2. Patients receive haploidentical stem cell transplantation.
3. Both patients and donors are CMV seropositive (IgG positive).
4. Subjects must be capable of, and willing to provide written informed consent to participate in the study. Subjects unable to provide written informed consent by themselves may be consented through their legal representative.

Exclusion Criteria:

1. Participation in another industry-sponsored clinical study where treatment for CMV is already specified by the study protocol.
2. Patients received other adoptive immunotherapy such as donor lymphocyte infusion (DLI), Epstein-Barr virus (EBV)-specific T cells and so on.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Virologic efficacy of CMVpp65-specific T cells for prophylaxis against refractory CMV infection after haploidentical stem cell transplantation | 6 months
  Virologic efficacy defined as reduction of refractory CMV infection during 6 months after transplantation
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 after adoptive transfer of CMV-specific T-cells | 6 months
  Patients were closely monitored for acute infusion-related toxicities during the first 2 to 4 hours following T-cell transfer and later on for acute and chronic GVHD during the whole observation period.

SECONDARY OUTCOMES:
Using Flow cytometry to evaluate the CMV-specific T cells reconstitution before and after CMV-CTL adoptive infusion post transplantation | 6 months
  Immunologic efficacy defined as in vivo reconstitution of CMV-specific antiviral immunity after adoptive transfer of CMV-CTLs
Reduction complications associated with CMV infection | 6 months
Reduction relapse rate of the primary disease | 6 months
Increase overall survival | 6 months
Increase disease-free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-jun Huang, MD,PHD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital & Peking University Institute of Hematology, Beijing Key Laboratory of Hematopoietic Stem Cell Transplantation, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao XY, Pei XY, Chang YJ, Yu XX, Xu LP, Wang Y, Zhang XH, Liu KY, Huang XJ. First-line Therapy With Donor-derived Human Cytomegalovirus (HCMV)-specific T Cells Reduces Persistent HCMV Infection by Promoting Antiviral Immunity After Allogenic Stem Cell Transplantation. Clin Infect Dis. 2020 Mar 17;70(7):1429-1437. doi: 10.1093/cid/ciz368. PMID 31067570